CLINICAL TRIAL: NCT00793468
Title: A Study to Investigate the Effects of GSK598809 in Newly Abstinent Nicotine-dependent Subjects.
Brief Title: Relapse Prevention Study in Newly Abstinent Smokers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prior to enrollment of patients
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 108428
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Substance Dependence
Keywords: nicotine dependence; smoking; pharmacological treatment; relapse prevention
MeSH Terms: conditions — Substance-Related Disorders; Tobacco Use Disorder; Smoking | interventions — GSK598809

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Subjects in placebo arm will be taking placebo once daily for 12 weeks from week 5 to 16.
  Interventions: Drug: GSK598809; Drug: Nicotine Replacement Transdermal Patch; Drug: Placebo
- GSK598809 Arm (Experimental): Subjects in GSK598809 arm will be taking GSK598809 once daily for 12 weeks from weeks 5 to 16.
  Interventions: Drug: GSK598809; Drug: Nicotine Replacement Transdermal Patch

INTERVENTIONS:
Drug: GSK598809 — GSK598809 once daily for 12 weeks
Drug: Nicotine Replacement Transdermal Patch — All subjects will be treated during the 4 week open-label smoking cessation phase of the study. During Weeks 1-3, subjects will receive 21mg/day, and during Week 4, subjects will receive 14 mg/day. Those subjects who reached continuous abstinence on at least week 4 of the open-label phase will receive 7mg/day during Week 5 while taking GSK598809 or placebo.
Drug: Placebo — Placebo once daily for 12 weeks
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to determine the effect of GSK598809 as compared to placebo in preventing recently-quit smokers from going back to smoking.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of GSK598809 compared to placebo for the prevention of relapse to smoking in recently abstinent smokers. Subjects who meet eligibility criteria will enter a 4-week open label treatment period during which they will receive nicotine replacement therapy (NRT). Subjects who have achieved at least one week of abstinence during the last week of an open label treatment period will be randomized to either GSK598809 or placebo in the double-blind treatment period and followed for another 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* has smoked at least 10 cigarettes a day for at least 2 years
* has had multiple previous attempts to quit smoking and relapsed to smoking.
* generally healthy

Exclusion Criteria:

* cannot be using smokeless tobacco of any type or has tried to quit with medicine.
* does not abuse alcohol or drugs
* certain emotional problems being treated with medications
* pregnant or breast feeding female

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Continuous smoking abstinence | weeks 13 through 16

SECONDARY OUTCOMES:
safety endpoints including vital signs, weight, ECGs, safety laboratory test and adverse events | weeks 1 through 16 and follow-up phase
Weekly point prevalence abstinence | Weeks 6, 8, 10, 12, 14, and 16
drug exposure level | weeks 6-16

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (10):
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas